CLINICAL TRIAL: NCT01092182
Title: Phase II Study of Dose-Adjusted EPOCH+/-Rituximab in Adults With Untreated Burkitt Lymphoma, c-MYC Positive Diffuse Large B-Cell Lymphoma and Plasmablastic Lymphoma
Brief Title: Phase II Study of Dose-Adjusted EPOCH-Rituximab in Adults With Untreated Burkitt Lymphoma and c-MYC+ Diffuse Large B-Cell Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Mark Roschewski, M.D., Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 100052; 10-C-0052
Record Dates: First submitted 2010-03-23; First posted 2010-03-24 (Estimated); Results first posted 2021-10-19 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Burkitt Lymphoma; Diffuse Large B-cell Lymphoma, c-MYC Positive; Plasmablastic Lymphoma
Keywords: Microarray; Toxicity; Therapeutic Index; HIV Positive; HIV Negative; HIV Infections
MeSH Terms: conditions — Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Plasmablastic Lymphoma; HIV Seropositivity; HIV Infections | interventions — Etoposide; Prednisone; Vincristine; Cyclophosphamide; Doxorubicin; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group A - Burkitt lymphoma Low Risk Arm (Experimental): Burkitt lymphoma Low Risk Arm Etoposide, prednisone, vincristine, cyclophosphamide, doxorubicin, and rituximab (EPOCH-R) every 21 days for 6 cycles
  Interventions: Drug: EPOCH-RR
- Group B - Burkitt lymphoma High Risk Arm (Experimental): Burkitt lymphoma High Risk Arm Etoposide, prednisone, vincristine, cyclophosphamide, doxorubicin, and rituximab (EPOCH-R) every 21 days for 6 cycles
  Interventions: Drug: EPOCH-R
- Group C - DLBCL high risk arm (Experimental): Diffuse large B-cell lymphoma (DLBCL) high risk arm Etoposide, prednisone, vincristine, cyclophosphamide, doxorubicin, and rituximab (EPOCH-R) every 21 days for 6 cycles
  Interventions: Drug: EPOCH-R

INTERVENTIONS:
Drug: EPOCH-R — Etoposide, prednisone, vincristine, cyclophosphamide, doxorubicin, and rituximab (EPOCH-R) every 21 days for 6 cycles
  Other Names: Etoposide; Prednisone; Vincristine; Cyclophosphamide; Doxorubicin; Rituximab
  Arms: Group B - Burkitt lymphoma High Risk Arm; Group C - DLBCL high risk arm
Drug: EPOCH-RR — Etoposide, prednisone, vincristine, cyclophosphamide, doxorubicin, and rituximab (EPOCH-R) every 21 days for 3 cycles
  Other Names: Etoposide; Prednisone; Vincristine; Cyclophosphamide; Doxorubicin; Rituximab
  Arms: Group A - Burkitt lymphoma Low Risk Arm

SUMMARY:
Background:

* Burkitt lymphoma/leukemia (BL) is highly treatable, but most of the standard therapies require multiple doses of intensive chemotherapy that may require long hospital stays and frequently have severe side effects. In addition, BL is a fairly common type of cancer in patients who also have human immunodeficiency virus (HIV), but treatment outcomes are poor because standard treatments do not work very well in HIV-positive patients and the more intense treatment regimens are highly toxic. New approaches are needed that expand the ways to treat BL with the same efficiency but with reduced side effects.
* Etoposide, prednisone, vincristine, cyclophosphamide, doxorubicin, and rituximab (DA-EPOCH-R) is a standard chemotherapy treatment that consists of the drugs etoposide, prednisone, vincristine, cyclophosphamide, doxorubicin, and rituximab. It may be able to treat BL with similar effectiveness but with fewer side effects. Researchers are interested in confirming the results of previous studies that investigated the effectiveness of DA-EPOCH-R in treating BL.

Objectives:

- To determine the safety and effectiveness of DA-EPOCH-R in treating Burkitt lymphoma.

Eligibility:

- Individuals at least 18 years of age who have been diagnosed with Burkitt lymphoma and have not had any prior chemotherapy treatments.

Design:

* Individuals will have a series of blood and other tests to determine their suitability for participating in the study. Eligible participants will be divided into high-risk and low-risk groups based on their disease prognosis and the possibility that the BL may or already has spread into the central nervous system.
* Participants will receive intravenous infusion of the six chemotherapy drugs in DA-EPOCH-R in 21-day treatment cycles. The exact doses will be adjusted depending on participants white blood cell counts and other tests.
* High-risk participants will receive six cycles of DA-EPOCH-R. To treat BL that may have entered the central nervous system, high-risk participants will also receive infusions of other chemotherapy drugs into their spinal fluid.
* Low-risk participants will receive up to six cycles of DA-EPOCH-R, with an additional dose of rituximab during each cycle.
* Frequent blood and urine tests will be performed during treatment, as well as body imaging scans and other tests of cancer progression as directed by the study doctors. Participants will receive additional medicines to help prevent possible adverse side effects of DA-EPOCH-R.
* Participants who respond successfully to the treatment will be asked to return for follow-up exams every 3 months for the first 18 months, then every year for the next 3 years. Participants who do not respond successfully to the treatment will be given the opportunity to participate in additional research and treatment protocols, if any are available.

DETAILED DESCRIPTION:
Background:

* Burkitt lymphoma/leukemia (BL) is highly curable. Standard treatment employs dose intense multi-agent chemotherapy and though effective is associated with high morbidity. Therefore, novel approaches are needed that improve the therapeutic index of BL while maintaining or improving efficacy. In human immunodeficiency virus (HIV)+ BL, outcome has been poor, mainly due to the use of cyclophosphamide, doxorubicin hydrochloride (hydroxydaunorubicin), vincristine sulfate (Oncovin), and prednisone (CHOP) based regimens in this disease.
* Two National Cancer Institute (NCI) phase II trials have used etoposide, prednisone, vincristine, cyclophosphamide, doxorubicin (EPOCH) chemotherapy with 1 or 2 doses of rituximab (R) per cycle in untreated BL. (Dose-adjusted) etoposide, prednisone, vincristine, cyclophosphamide, doxorubicin, and rituximab (DA-EPOCH)-Rituximab has been used in16 HIV negative BL, and 8 HIV positive patients have received 3 to 4 cycles of EPOCHRR to minimize toxicity and risk of opportunistic infections. All patients remain in continuous remission. Treatment was very well tolerated and represents a novel therapeutic strategy in BL.
* This trial seeks to assess the effectiveness of a risk adaptive approach with DA-EPOCHR in untreated BL (HIV+/-). Because this treatment represents a major conceptual departure from standard treatment, it is important to obtain additional Phase II results in limited/advanced stage BL
* c-MYC positive Diffuse large B cell (DLBCL) is a rare variant of Diffuse Large B-Cell Lymphoma (DLBCL). There is very little data on the biology of this disease and what the optimal therapeutic approach should be has not been defined. Therefore, based on our impression that this behaves aggressively and is likely characterized by a high tumor proliferation rate, we plan to accrue patients with this disease in addition to BL patients.
* Plasmablastic lymphoma, another variant of DLBCL is frequently characterized by the activation of MYC and has had a poor outcome historically with standard treatment. We plan to include these patients in the study also. As they are cluster of differentiation 20 (CD20) negative, they will receive DA-EPOCH without Rituximab.

Objectives:

* Determine progression free survival (PFS), event free survival (EFS) and overall survival (OS) of risk adaptive DA-EPOCH-R in untreated BL and c-MYC + DLBCL and DA-EPOCH in c-MYC+ plasmablastic lymphoma.
* Assess predictive value of early fluorodeoxyglucose (FDG)-positron emission tomography (PET)/computed tomography (CT) scans on PFS.
* Obtain pilot comparative molecular profiling in HIV negative and positive BL and c- MYC + DLBCL, including c-MYC+ plasmablastic lymphoma.

Eligibility:

* Burkitt lymphoma, c-MYC + DLBCL and c-MYC + plasmablastic lymphoma age greater than or equal to 18 years.
* No prior treatment except limited-field radiotherapy, short course of glucocorticoids and/or cyclophosphamide for an urgent problem at diagnosis.
* Adequate major organ function unless impairment due to lymphoma.

Study Design:

* Phase II Study of risk adapted DA-EPOCH-R in BL, c-MYC + DLBCL and DA-EPOCH in c-MYC+ plasmablastic lymphoma
* Low risk: DA-EPOCH-RR x 3 cycles.
* High risk , c-MYC + DLBCL and c-MYC+ plasmablastic lymphoma : DA-EPOCH (+/-) R x 6 cycles or 8 cycles in select patients.
* Cerebrospinal fluid (CSF) cytology and flow cytometry for analysis of BL.
* High Risk CSF negative - Prophylactic intrathecal treatment
* CSF positive - Active intrathecal treatment
* FDG-PET/CT pre- and post-cycle 2 in all patients.
* A total of 194 patients will be enrolled in the protocol.

ELIGIBILITY:
* INCLUSION CRITERIA:

Patients must have one of the following histologic diagnoses:

-Patients must have Burkitt Lymphoma. Effective with Amendment J (version date: 06/24/2014), the following histologies were removed as the maximum number allowed for these sub-groups has been reached: B-cell lymphoma: unclassifiable with features intermediate between Diffuse Large B cell lymphoma and Burkitt Lymphoma ; c-MYC + Diffuse large B-cell lymphoma (DLBCL) and c-MYC+ plasmablastic lymphoma.

If questions arise related to diagnosis, please contact the National Cancer Institute (NCI) Principal Investigator, Dr. Mark Roschewski or the NCI study coordinator, A. Nicole Lucas.

* Age greater than or equal to 18 years. Because no dosing or adverse event data are currently available on the use of etoposide, prednisone, vincristine, cyclophosphamide, doxorubicin, and rituximab (EPOCH-R) in patients <18 years of age, children are excluded from this study, but may be eligible for future pediatric trials
* Pathology confirmed by treating institutions Pathology Department.
* No prior treatment except patients may be entered if they have had prior limited-field radiotherapy, a short course of glucocorticoids, cyclophosphamide for an urgent problem at diagnosis (e.g. epidural cord compression, superior vena cava syndrome) and/or a single dose of intrathecal methotrexate (MTX) at the time of the pre-treatment diagnostic lumbar puncture.
* All disease stages.
* Human immunodeficiency virus (HIV) negative or positive.
* HIV positive patients on antiretroviral therapy regimen must be willing to suspend all Highly Active Antiretroviral Therapy (HAART) except in circumstances described in section 6.5.
* Eastern Cooperative Oncology Group (ECOG) 0-4
* Ability of patient or durable power of attorney (DPA) for healthcare to give informed consent.
* Hepatitis B + patients may be enrolled at the discretion of the investigator.

EXCLUSION CRITERIA:

* Patients with Primary central nervous system (CNS) Lymphoma.
* Inadequate renal function, defined as serum creatinine (Cr) > 1.5 or creatinine clearance < 50ml/min/1.73m^2 unless lymphoma related.
* Inadequate hepatic or hematological function: as follows, unless lymphoma-/disease-related: bilirubin greater than 2 mg/dl (total) except greater than 5 mg/dl in patients with Gilbert's syndrome as defined by greater than 80% unconjugated, absolute neutrophil count (ANC) less than 1000 and platelets less than 75,000.
* The effects of EPOCH-R on the developing human fetus are unknown. For this reason and because chemotherapy agents are known to be teratogenic, female subject of child-bearing potential not willing to use an acceptable method of birth control(i.e., a hormonal contraceptive, intra-uterine device, diaphragm with spermicide, condom with spermicide, or abstinence) for the duration of the study and one year beyond treatment completion will not be eligible to participate in the study.
* Female subject pregnant or breast-feeding. Confirmation that the subject is not pregnant must be established by a negative serum beta-human chorionic gonadotropin (beta-human chorionic gonadotropin (hCG) pregnancy test result obtained during screening. Pregnancy testing is not required for women without child-bearing potential.
* The effects of EPOCH-R on the developing human fetus are unknown. For this reason and because chemotherapy agents are known to be teratogenic, male subject unwilling to use an acceptable method for contraception for the duration of the study and one year beyond treatment completion, will not be eligible to participate in the study.
* History of a prior invasive malignancy in past 5 years.
* Active symptomatic ischemic heart disease, myocardial infarction or congestive heart failure within the past year. If echo is obtained the left ventricular ejection fraction (LVEF) should exceed 40%.
* Serious concomitant medical illnesses that would jeopardize the patient's ability to receive the regimen with reasonable safety.
* HIV positive patients with advanced immune suppression and evidence of HIV resistant to all combinations of antiretroviral therapy considered at high risk of non lymphoma related death within 12-months due to other acquired immunodeficiency syndrome (AIDS) complications should not be enrolled on the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 194 (Actual)
Dates: Start 2010-03-25 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2023-02-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark J Roschewski, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (30):
- United States (30):
  - UC San Diego Moores Cancer Center, La Jolla, California
  - UCLA Center for Clinical AIDS Research and Education, Los Angeles, California
  - Emory University /Winship Cancer Institute, Atlanta, Georgia
  - University of Illinois, Chicago, Illinois
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - University of Kentucky /Markey Cancer Center, Lexington, Kentucky
  - National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland
  - Massachusetts General Hospital Cancer Centers, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Fairview - Southdale Hospital, Edina, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Mount Sinai Hospital, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of Rochester, Rochester, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - Vidant Oncology-Kinston, Kinston, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Case Western Reserve University, Cleveland, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - University of Tennessee - Knoxville, Knoxville, Tennessee
  - UT Southwestern /Simmons Cancer Center- Dallas, Dallas, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
  - Froedtert and the Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data (IPD) recorded in the medical record will be shared with intramural investigators upon request. All collected IPD will be shared with collaborators under the terms of collaborative agreements.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely.
Access Criteria: Clinical data will be made available upon request to the study principal investigator.

REFERENCES:
- [Derived] Roschewski M, Dunleavy K, Abramson JS, Powell BL, Link BK, Patel P, Bierman PJ, Jagadeesh D, Mitsuyasu RT, Peace D, Watson PR, Hanna WT, Melani C, Lucas AN, Steinberg SM, Pittaluga S, Jaffe ES, Friedberg JW, Kahl BS, Little RF, Bartlett NL, Fanale MA, Noy A, Wilson WH. Multicenter Study of Risk-Adapted Therapy With Dose-Adjusted EPOCH-R in Adults With Untreated Burkitt Lymphoma. J Clin Oncol. 2020 Aug 1;38(22):2519-2529. doi: 10.1200/JCO.20.00303. Epub 2020 May 26. PMID 32453640
- [Derived] Dunleavy K, Fanale MA, Abramson JS, Noy A, Caimi PF, Pittaluga S, Parekh S, Lacasce A, Hayslip JW, Jagadeesh D, Nagpal S, Lechowicz MJ, Gaur R, Lucas A, Melani C, Roschewski M, Steinberg SM, Jaffe ES, Kahl B, Friedberg JW, Little RF, Bartlett NL, Wilson WH. Dose-adjusted EPOCH-R (etoposide, prednisone, vincristine, cyclophosphamide, doxorubicin, and rituximab) in untreated aggressive diffuse large B-cell lymphoma with MYC rearrangement: a prospective, multicentre, single-arm phase 2 study. Lancet Haematol. 2018 Dec;5(12):e609-e617. doi: 10.1016/S2352-3026(18)30177-7. PMID 30501868
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2010-C-0052.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Low-risk Burkitt Lymphoma (BL): Burkitt lymphoma Low Risk Arm
  Etoposide, prednisone, vincristine, cyclophosphamide, doxorubicin, and rituximab (EPOCH-R) every 21 days for 6 cycles
- High-Risk Burkitt Lymphoma (BL): Burkitt lymphoma High Risk Arm
  Etoposide, prednisone, vincristine, cyclophosphamide, doxorubicin, and rituximab (EPOCH-R) every 21 days for 6 cycles
- High-Risk Diffuse Large B Cell Lymphoma (DLBCL): High-Risk Diffuse Large B Cell Lymphoma
  Etoposide, prednisone, vincristine, cyclophosphamide, doxorubicin, and rituximab (EPOCH-R) every 21 days for 6 cycles
Period: Overall Study
Arm/Group | Low-risk Burkitt Lymphoma (BL) | High-Risk Burkitt Lymphoma (BL) | High-Risk Diffuse Large B Cell Lymphoma (DLBCL)
Started | 15 | 98 | 81
Completed | 14 | 80 | 53
Not Completed | 1 | 18 | 28
Not completed — Death | 0 | 5 | 3
Not completed — participant safety | 1 | 2 | 0
Not completed — Physician Decision | 0 | 6 | 0
Not completed — Did not meet criteria | 0 | 0 | 25
Not completed — Non-compliance | 0 | 3 | 0
Not completed — Participant refused follow-up | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Group A - Low-risk Burkitt Lymphoma (BL): Burkitt lymphoma Low Risk Arm
  Etoposide, prednisone, vincristine, cyclophosphamide, doxorubicin, and rituximab (EPOCH-R) every 21 days for 6 cycles
- Group B - High-Risk Burkitt Lymphoma (BL): Burkitt lymphoma High Risk Arm
  Etoposide, prednisone, vincristine, cyclophosphamide, doxorubicin, and rituximab (EPOCH-R) every 21 days for 6 cycles
- Group C - High-Risk Diffuse Large B Cell Lymphoma (DLBCL): Diffuse large B-cell lymphoma (DLBCL) high risk arm
  Etoposide, prednisone, vincristine, cyclophosphamide, doxorubicin, and rituximab (EPOCH-R) every 21 days for 6 cycles
- Total: Total of all reporting groups
Arm/Group | Group A - Low-risk Burkitt Lymphoma (BL) | Group B - High-Risk Burkitt Lymphoma (BL) | Group C - High-Risk Diffuse Large B Cell Lymphoma (DLBCL) | Total
Number analyzed (Participants) | 15 | 98 | 81 | 194
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 13 | 84 | 55 | 152
  >=65 years | 2 | 14 | 26 | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.47 (14.85) | 46.35 (17.53) | 57.47 (14) | 51.39 (16.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 20 | 20 | 44
  Male | 11 | 78 | 61 | 150
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 2 | 16 | 6 | 24
  White | 11 | 65 | 66 | 142
  Indian or Alaska Native | 1 | 0 | 0 | 1
  Indian or Alaska Native + White | 0 | 1 | 0 | 1
  Asian | 1 | 5 | 2 | 8
  Race Unknown/Not Reported | 0 | 11 | 7 | 18
  Hispanic or Latino | 1 | 10 | 4 | 15
  Not Hispanic or Latino | 14 | 80 | 72 | 166
  Ethnicity Unknown/Not Reported | 0 | 8 | 5 | 13
Region of Enrollment [Number; unit: participants]
  United States | 15 | 98 | 81 | 194
Eastern Cooperative Oncology Group (ECOG) [Count of Participants; unit: Participants] — ECOG Criteria:
  0 - Normal activity
  1. - Symptoms, but ambulatory.
  2. - In bed <50% of the time.
  3. - In bed >50% of the time.
  4. - 100% bedridden.
  Participants
    0 | 11 | 39 | 26 | 76
    1 | 4 | 38 | 37 | 79
    2 | 0 | 14 | 9 | 23
    3 | 0 | 4 | 7 | 11
    4 | 0 | 3 | 2 | 5
Baseline Risk Stratification [Count of Participants; unit: Participants] — Low Risk disease High Risk disease
  Participants
    Low Risk | 15 | 0 | 0 | 15
    High Risk | 0 | 98 | 81 | 179
International Prognostic Index Score 0-5 [Count of Participants; unit: Participants] — International Prognostic Index Score 0 -1 is low risk 2 is low-intermediate risk 3 is high-intermediate risk 4 - 5 is high risk
  Participants
    0 | 12 | 8 | 7 | 27
    1 | 3 | 19 | 7 | 29
    2 | 0 | 20 | 28 | 48
    3 | 0 | 24 | 30 | 54
    4 | 0 | 24 | 5 | 29
    5 | 0 | 3 | 4 | 7
Histology [Count of Participants; unit: Participants]
  High Grade B Cell Lymphoma Double-hit (HGBL DH) | NA — This study specific measure is only applicable to Group C. | NA — This study specific measure is only applicable to Group C. | 24 | NA — Total not calculated because data are not available (NA) in one or more arms.
  High Grade B Cell Lymphoma Not Otherwise Specified (HGBL NOS) | NA — This study specific measure is only applicable to Group C. | NA — This study specific measure is only applicable to Group C. | 12 | NA — Total not calculated because data are not available (NA) in one or more arms.
  Diffuse Large B-Cell Lymphoma (DLBCL) | NA — This study specific measure is only applicable to Group C. | NA — This study specific measure is only applicable to Group C. | 44 | NA — Total not calculated because data are not available (NA) in one or more arms.
  Plasmablastic | NA — This study specific measure is only applicable to Group C. | NA — This study specific measure is only applicable to Group C. | 1 | NA — Total not calculated because data are not available (NA) in one or more arms.

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Kaplan-Meier Curve Progression Free Survival (PFS) Constructed With an 95% Confidence Interval
Description: PFS is the time interval from start of treatment to documented evidence of disease progression. Disease progression was measured by the International Workshop Criteria (IWC). Progression is a positive positron emission tomography (PET) finding corresponding to the computed tomography (CT) abnormality (new lesion, increasing size of previous lesion), or a negative PET and a CT abnormality (new lesion, increasing size of previous lesion) of < 1.5 cm (< 1.0 cm in the lungs). Kaplan-Meier curves were constructed with an 95% confidence interval.
Time Frame: Time of progression or death at 4 years
Population: Those participants that were not analyzed for PFS were screen failures (did not have MYC+ Diffuse Large B-Cell Lymphoma (DLBCL).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group A - Low-risk Burkitt Lymphoma (BL) | Group B - High-Risk Burkitt Lymphoma (BL) | Group C - High-Risk Diffuse Large B Cell Lymphoma (DLBCL)
Number analyzed (Participants) | 15 | 98 | 53
percentage of participants | 100 [1 to 100] | 82.1 [72.7 to 88.5] | 71.0 [56.5 to 81.4]

2. Primary Outcome: Percentage of Participants With Kaplan-Meier Curve Event Free Survival (EFS) Constructed With an 95% Confidence Interval
Description: EFS was determined from the date of enrolment in the study until the date of progression, last documentation of disease at or after the last treatment cycle, death, or last follow-up (whichever occurred first). Disease progression was measured by the International Workshop Criteria (IWC). Progression is a positive positron emission tomography (PET) finding corresponding to the computed tomography (CT) abnormality (new lesion, increasing size of previous lesion), or a negative PET and a CT abnormality (new lesion, increasing size of previous lesion) of < 1.5 cm (< 1.0 cm in the lungs). Kaplan-Meier curves were constructed with an 95% confidence interval.
Time Frame: At 4 years
Population: Those participants that were not analyzed for EFS were screen failures (did not have MYC+ Diffuse Large B-Cell Lymphoma (DLBCL).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group A - Low-risk Burkitt Lymphoma (BL) | Group B - High-Risk Burkitt Lymphoma (BL) | Group C - High-Risk Diffuse Large B Cell Lymphoma (DLBCL)
Number analyzed (Participants) | 15 | 98 | 53
percentage of participants | 100 [1 to 100] | 82.1 [72.7 to 88.5] | 71.0 [58.5 to 81.4]

3. Primary Outcome: Percentage of Participants Kaplan-Meier Curve Overall Survival (OS) Constructed With an 95% Confidence Interval
Description: OS was calculated from the enrolment date until date of death or last follow-up using the Kaplan Meier. Kaplan-Meier curves were constructed with an 95% confidence interval.
Time Frame: At 4 years
Population: Those participants that were not analyzed for OS were screen failures (did not have MYC+ Diffuse Large B-Cell Lymphoma (DLBCL).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group A - Low-risk Burkitt Lymphoma (BL) | Group B - High-Risk Burkitt Lymphoma (BL) | Group C - High-Risk Diffuse Large B Cell Lymphoma (DLBCL)
Number analyzed (Participants) | 15 | 98 | 53
percentage of participants | 100 [1 to 100] | 84.9 [75.8 to 90.8] | 76.7 [62.6 to 86.1]

4. Secondary Outcome: Kaplan-Meier Progression Free Survival (PFS) Constructed With an 95% Confidence Interval in Participants Who Underwent Fluorodeoxyglucose (FDG)-Positron Emission Tomography (PET) and/or Computed Tomography (CT) Scans After Cycle 2
Description: The predictive value of early FDG-PET/CT scans on PFS was assessed after cycle 2. PFS is the time interval from start of treatment to documented evidence of disease progression, assessed by the International Workshop Criteria (IWC). Progression is a positive positron emission tomography (PET) finding corresponding to the computed tomography (CT) abnormality (new lesion, increasing size of previous lesion), or a negative PET and a CT abnormality (new lesion, increasing size of previous lesion) of < 1.5 cm (< 1.0 cm in the lungs). Kaplan-Meier curves were constructed with an 95% confidence interval.
Time Frame: After 2 cycles of therapy and prior to cycle 3
Population: 51/98 participants and 34/81 participants did not receive a PET scan.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group A - Low-risk Burkitt Lymphoma (BL) | Group B - High-Risk Burkitt Lymphoma (BL) | Group C - High-Risk Diffuse Large B Cell Lymphoma (DLBCL)
Number analyzed (Participants) | 15 | 51 | 34
percentage of participants | 100 [1 to 100] | 90.0 [77.7 to 95.7] | 78.7 [60.5 to 89.2]

5. Other Pre Specified Outcome: Number of Participants With Serious and Non-serious Adverse Events Assessed by the Common Terminology Criteria for Adverse Events (CTCAE v4.0)
Description: Here is the number of participants with serious and non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v4.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Date treatment consent signed to date off study, approximately 102 months and 25 days for Group A, 125 months and 28 days for Group B and 117 months and 29 days for group C.
Measure: Count of Participants; unit: Participants
Arm/Group | Group A - Low-risk Burkitt Lymphoma (BL) | Group B - High-Risk Burkitt Lymphoma (BL) | Group C - High-Risk Diffuse Large B Cell Lymphoma (DLBCL)
Number analyzed (Participants) | 15 | 98 | 81
Participants | 13 | 87 | 72

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, approximately 102 months and 25 days for Group A, 125 months and 28 days for Group B and 117 months and 29 days for group C.
Arm/Group | Group A - Low-risk Burkitt Lymphoma (BL) | Group B - High-Risk Burkitt Lymphoma (BL) | Group C - High-Risk Diffuse Large B Cell Lymphoma (DLBCL)
All-Cause Mortality (participants affected / at risk) | 0/15 | 16/98 | 3/81
Serious Adverse Events (participants affected / at risk) | 3/15 | 58/98 | 33/81
Other Adverse Events (participants affected / at risk) | 13/15 | 88/98 | 71/81
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A - Low-risk Burkitt Lymphoma (BL) (N=15) | Group B - High-Risk Burkitt Lymphoma (BL) (N=98) | Group C - High-Risk Diffuse Large B Cell Lymphoma (DLBCL) (N=81)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (3) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 3 (4)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (2) | 12 (21) | 4 (5)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiac disorders - Other, hypotension (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Catheter related infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Cerebrospinal fluid leakage (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Chest pain - cardiac (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1)
Death NOS (General disorders) | 0 (0) | 10 (10) | 9 (9)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 3 (3) | 2 (2)
Device related infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (3)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Edema limbs (General disorders) | 0 (0) | 1 (1) | 0 (0)
Ejection fraction decreased (Investigations) | 0 (0) | 1 (1) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 27 (48) | 11 (16)
Fever (General disorders) | 0 (0) | 6 (7) | 1 (1)
Gastric perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal disorders - Other, bleeding (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1)
General disorders and administration site conditions - Other, specify (General disorders) | 0 (0) | 1 (1) | 0 (0) — Weakness, difficulty swallowing, esophagitis
Hallucinations (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Hematoma (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Hematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 2 (2)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (3)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 3 (3) | 2 (2)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 4 (5) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Infections and infestations - Other, cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Infusion related reaction (General disorders) | 0 (0) | 1 (1) | 0 (0)
Intracranial hemorrhage (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Jejunal perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1)
Lung infection (Infections and infestations) | 0 (0) | 3 (3) | 1 (1)
Lymphocyte count decreased (Investigations) | 1 (1) | 7 (14) | 3 (7)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 8 (11) | 0 (0)
Multi-organ failure (General disorders) | 0 (0) | 1 (1) | 2 (2)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 2 (3)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) — Cholangiocarcinoma of liver
Neutrophil count decreased (Investigations) | 1 (1) | 11 (26) | 5 (8)
Oral pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Phlebitis infective (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 6 (12) | 4 (6)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Renal and urinary disorders - Other, acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 3 (3)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) — Pharyngeal pain
Restrictive cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 6 (6) | 4 (6)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 4 (4)
Thromboembolic event (Vascular disorders) | 0 (0) | 3 (3) | 1 (1)
Toxic epidermal necrolysis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Treatment related secondary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Tumor lysis syndrome (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Vascular access complication (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0)
Vasovagal reaction (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 3 (3) | 2 (3)
White blood cell decreased (Investigations) | 0 (0) | 15 (38) | 5 (7)
Gastrointestinal disorders - Other, heme positive stool (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal disorders - Other, odynohagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Infections and infestations - Other, clostridium difficile (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Infections and infestations - Other, influenza A/H1N1 (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Infections and infestations - Other, Infected Cholecystostomy tube in setting of neutropenia? (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Infections and infestations - Other, neutropenic fever (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Infections and infestations - Other, liver infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1) — Progressive disease
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A - Low-risk Burkitt Lymphoma (BL) (N=15) | Group B - High-Risk Burkitt Lymphoma (BL) (N=98) | Group C - High-Risk Diffuse Large B Cell Lymphoma (DLBCL) (N=81)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0)
Abdominal infection (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 8 (11) | 5 (5)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 0 (0) | 2 (2)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 2 (2) | 1 (1)
Alanine aminotransferase increased (Investigations) | 2 (2) | 15 (23) | 7 (14)
Alkaline phosphatase increased (Investigations) | 0 (0) | 7 (10) | 12 (21)
Alkalosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Allergic reaction (Immune system disorders) | 0 (0) | 3 (3) | 2 (2)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 4 (6) | 9 (14) | 6 (6)
Anal fistula (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 6 (9) | 62 (216) | 53 (181)
Anorectal infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 9 (10) | 6 (7)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 13 (18) | 7 (12)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 3 (3)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 5 (6) | 2 (2)
Atrial flutter (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 7 (10) | 7 (7)
Bladder infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Bloating (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Blood and lymphatic system disorders - Other, DVT (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 2 (2) | 9 (13) | 5 (9)
Blurred vision (Eye disorders) | 0 (0) | 3 (3) | 2 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (3) | 9 (13) | 7 (10)
Bronchial infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
CD4 lymphocytes decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Cardiac disorders - Other, 23% decreased EF (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiac troponin I increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Cardiac troponin T increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Catheter related infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Cerebrospinal fluid leakage (Nervous system disorders) | 0 (0) | 2 (3) | 0 (0)
Chest pain - cardiac (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Chills (General disorders) | 1 (1) | 5 (6) | 2 (2)
Cognitive disturbance (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Confusion (Psychiatric disorders) | 0 (0) | 3 (3) | 2 (2)
Constipation (Gastrointestinal disorders) | 6 (6) | 20 (23) | 22 (37)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 6 (6) | 1 (1)
Creatinine increased (Investigations) | 0 (0) | 1 (1) | 1 (1)
Death NOS (General disorders) | 0 (0) | 2 (2) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 7 (11) | 2 (3)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1)
Delusions (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 3 (3) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 18 (20) | 17 (22)
Dizziness (Nervous system disorders) | 0 (0) | 7 (9) | 3 (5)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1) | 5 (6)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 2 (3) | 3 (3)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 4 (4) | 2 (2)
Dysphasia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 8 (9) | 7 (9)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 2 (2)
Edema limbs (General disorders) | 0 (0) | 3 (3) | 11 (12)
Elevated LFT's (Investigations) | 0 (0) | 1 (1) | 0 (0)
Elevated bilirubin (Investigations) | 0 (0) | 1 (1) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Enterocolitis infectious (Infections and infestations) | 0 (0) | 2 (2) | 4 (4)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Esophageal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Esophageal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Esophagitis (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Eye infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Eyelid function disorder (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Facial nerve disorder (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 1 (1)
Fatigue (General disorders) | 4 (7) | 22 (28) | 22 (35)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 29 (42) | 22 (35)
Fecal incontinence (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Fever (General disorders) | 1 (1) | 13 (16) | 8 (10)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2)
Floaters (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Flu like symptoms (General disorders) | 0 (0) | 1 (1) | 2 (2)
GGT increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Gait disturbance (General disorders) | 0 (0) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 2 (2) | 2 (2)
Gastrointestinal disorders - Other, epigastric pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
General disorders and administration site conditions - Other, cerebellar infarct (General disorders) | 0 (0) | 2 (3) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (7) | 5 (6)
Glucose intolerance (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (2) | 25 (31) | 11 (13)
Hematoma (Vascular disorders) | 0 (0) | 3 (4) | 0 (0)
Hematuria (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0)
Hemorrhoids (Gastrointestinal disorders) | 0 (0) | 3 (3) | 1 (2)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 0 (0)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 1 (1)
Hot flashes (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 3 (3)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 16 (42) | 15 (37)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3) | 3 (3)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 3 (4)
Hypernatremia (Metabolism and nutrition disorders) | 0 (0) | 4 (5) | 8 (17)
Hypertension (Vascular disorders) | 1 (1) | 5 (9) | 6 (12)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperuricemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 2 (2)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 18 (32) | 15 (27)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 17 (32) | 17 (28)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 4 (7) | 3 (3)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 21 (32) | 18 (36)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 7 (13) | 6 (16)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 14 (19) | 6 (8)
Hypophosphatemia (Metabolism and nutrition disorders) | 2 (2) | 22 (36) | 20 (29)
Hypotension (Vascular disorders) | 0 (0) | 8 (9) | 6 (8)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 3 (4)
Infections and infestations - Other, bacteremia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Infusion related reaction (General disorders) | 0 (0) | 2 (2) | 3 (3)
Insomnia (Psychiatric disorders) | 1 (1) | 10 (12) | 6 (6)
Investigations - Other, disease progression (Investigations) | 0 (0) | 0 (0) | 1 (1)
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Laryngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 3 (3) | 2 (2)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Lymphocyte count decreased (Investigations) | 5 (11) | 54 (277) | 49 (239)
Lymphocyte count increased (Investigations) | 0 (0) | 1 (1) | 3 (3)
Memory impairment (Nervous system disorders) | 0 (0) | 2 (5) | 1 (1)
Metabolism and nutrition disorders - Other, elevated LDH (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Movements involuntary (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Mucosal infection (Infections and infestations) | 0 (0) | 8 (12) | 4 (5)
Mucositis oral (Gastrointestinal disorders) | 1 (1) | 23 (47) | 20 (31)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0)
Muscle weakness trunk (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) — PICC line-associated shoulder pain
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (2)
Nail discoloration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Nail loss (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (3) | 18 (25) | 11 (16)
Neck edema (General disorders) | 0 (0) | 2 (2) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3) | 1 (1)
Nervous system disorders - Other, numbness in left arm (Nervous system disorders) | 1 (3) | 0 (0) | 2 (6)
Neutrophil count decreased (Investigations) | 5 (6) | 55 (201) | 49 (178)
Non-cardiac chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Oral hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Oral pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (5)
Pain (General disorders) | 1 (1) | 10 (14) | 6 (7)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3) | 3 (4)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Pancreatic enzymes decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Papulopustular rash (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Paresthesia (Nervous system disorders) | 0 (0) | 5 (5) | 3 (10)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 8 (9) | 8 (9)
Peripheral sensory neuropathy (Nervous system disorders) | 5 (5) | 26 (33) | 22 (25)
Peritoneal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Personality change (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Pharyngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Photophobia (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 3 (3) | 52 (161) | 43 (159)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 2 (4) | 2 (2)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3) | 1 (1)
Psychiatric disorders - Other, non verbal (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 3 (3)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Rash pustular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Rectal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Renal and urinary disorders - Other, dysuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Retinal detachment (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Rhinitis infective (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Scrotal pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 2 (2)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 2 (2) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 4 (4) | 4 (5)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Skin and subcutaneous tissue disorders - Other, abdominal abscess (Skin and subcutaneous tissue disorders) | 2 (2) | 4 (5) | 1 (1)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (5) | 1 (1)
Stomach pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Superficial thrombophlebitis (Vascular disorders) | 0 (0) | 2 (2) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 5 (7) | 2 (2)
Thromboembolic event (Vascular disorders) | 0 (0) | 6 (6) | 5 (5)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0)
Tracheal fistula (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Tumor lysis syndrome (Metabolism and nutrition disorders) | 0 (0) | 4 (4) | 0 (0)
Typhlitis (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Upper respiratory infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Urethral infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2)
Urinary tract infection (Infections and infestations) | 0 (0) | 8 (9) | 8 (11)
Urinary tract pain (Renal and urinary disorders) | 1 (1) | 1 (1) | 2 (2)
Urinary urgency (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Urine output decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 9 (14) | 7 (8)
Watering eyes (Eye disorders) | 0 (0) | 0 (0) | 2 (2)
Weight gain (Investigations) | 0 (0) | 3 (5) | 1 (1)
Weight loss (Investigations) | 0 (0) | 2 (2) | 5 (8)
White blood cell decreased (Investigations) | 7 (10) | 47 (212) | 52 (218)
Wound infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Blood and lymphatic system disorders - Other, leukopenia (Blood and lymphatic system disorders) | 0 (0) | 2 (4) | 0 (0)
Blood and lymphatic system disorders - Other, low ANC (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Blood and lymphatic system disorders - Other, low platelet count (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0)
Blood and lymphatic system disorders - Other, T bili (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2)
Blood and lymphatic system disorders - Other, thrombosis/embolism (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
General disorders and administration site conditions - Other, sacral pressure ulcer (General disorders) | 0 (0) | 1 (1) | 0 (0)
General disorders and administration site conditions - Other, thalmic infarct (General disorders) | 0 (0) | 1 (1) | 0 (0)
Infections and infestations - Other, Blood (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Infections and infestations - Other, blood infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Infections and infestations - Other, blood, E. coli (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Infections and infestations - Other, bacteremia, Klebsiella infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Infections and infestations - Other, candida oral infection (Infections and infestations) | 0 (0) | 1 (2) | 0 (0)
Infections and infestations - Other, clostridium difficile (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Infections and infestations - Other, CMV reactivation (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Infections and infestations - Other, encephalitis, persistent (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Infections and infestations - Other, gastrointestinal tract (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Infections and infestations - Other, infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Infections and infestations - Other, infection-oral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Infections and infestations - Other, L posterior lung (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Infections and infestations - Other, left orbital cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Infections and infestations - Other, MRSA (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Infections and infestations - Other, oral cavity (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Infections and infestations - Other, parasitic infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Infections and infestations - Other, PICC line infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Infections and infestations - Other, polymicrobial bacteremia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Infections and infestations - Other, throat (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Infections and infestations - Other, thrush (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Infections and infestations - Other, VRE (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Infections and infestations - Other, VRE-blood stream (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Infections and infestations - Other, blood, candida glabrata (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Infections and infestations - Other, herpes simplex oral ulcer (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Infections and infestations - Other, oral thrush (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Investigations - Other, heartburn (Investigations) | 0 (0) | 1 (1) | 0 (0)
Investigations - Other, night sweats (Investigations) | 0 (0) | 1 (1) | 0 (0)
Investigations - Other, fluid overload (Investigations) | 0 (0) | 1 (1) | 0 (0)
Metabolism and nutrition disorders - Other, malnutrition (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal and connective tissue disorder - Other, shin pain with numbness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Nervous system disorders - Other, neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 1 (5)
Nervous system disorders - Other, neuropathy, upper bilateral extremities (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Skin and subcutaneous tissue disorders - Other, blister ball of R foot (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other, dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Skin and subcutaneous tissue disorders - Other, forehead itching (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other, skin darkening (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Skin and subcutaneous tissue disorders - Other, vitiligo (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Skin and subcutaneous tissue disorders - Other, pressure ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other, scalp wound (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-09-20): https://cdn.clinicaltrials.gov/large-docs/82/NCT01092182/Prot_SAP_000.pdf
  • Informed Consent Form (2019-12-03): https://cdn.clinicaltrials.gov/large-docs/82/NCT01092182/ICF_001.pdf